CLINICAL TRIAL: NCT05851404
Title: Management of Indeterminate Thyroid Nodules Across Different World Regions: a Multicentric International Study
Brief Title: Management of Indeterminate Thyroid Nodules Across Different World Regions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Fabio Medas, Associate Professor, University of Cagliari
Other Study IDs: UNICA-MEDAS-23-01
Record Dates: First submitted 2023-05-01; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Indeterminate Thyroid Nodules
Keywords: Indeterminate thyroid nodule; Thyroid carcinoma
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Thyroidectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- South East Asian Region (SEAR): Patients that underwent thyroidectomy for indeterminate thyroid nodules in the SEAR
  Interventions: Procedure: Thyroidectomy
- Americas Region (AMR): Patients that underwent thyroidectomy for indeterminate thyroid nodules in the AMR
  Interventions: Procedure: Thyroidectomy
- Eastern Mediterranean Region (EMR): Patients that underwent thyroidectomy for indeterminate thyroid nodules in the EMR
  Interventions: Procedure: Thyroidectomy
- the Europe Region (EUR): Patients that underwent thyroidectomy for indeterminate thyroid nodules in the EUR
  Interventions: Procedure: Thyroidectomy
- Western Pacific Region (WPR): Patients that underwent thyroidectomy for indeterminate thyroid nodules in the WPR
  Interventions: Procedure: Thyroidectomy

INTERVENTIONS:
Procedure: Thyroidectomy — Total thyroidectomy or lobectomy

SUMMARY:
Thyroid carcinoma (TC) is the most common endocrine malignancy, affecting 0.2-1.5% of individuals worldwide. The rising incidence rate of TC is mostly related to the expanding use of high-quality imaging techniques, with an increase in the detection of thyroid nodules. Fine needle aspiration cytology (FNAC) is the most accurate, rapid, safe, and cost-effective test for the evaluation of thyroid nodules, with high specificity and sensitivity. Nevertheless, FNAC is particularly unreliable in differentiating between benign and malignant nodules that fall under the category of indeterminate thyroid nodules (class III and class IV according to Bethesda Classification[2]). In fact, in these cases, the expected malignancy rates are 5-15% and 15-30%, respectively. Thus, most patients with indeterminate thyroid nodules undergo an operation that is indeed unnecessary, while representing a risk for surgical complications and a cost for health-care systems.

We aim to evaluate different approaches to indeterminate nodules across different countries in the world.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Bethesda III / Bethesda IV thyroid nodules

Exclusion Criteria:

* Patients with preoperative diagnosis of lymph node metastases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We aim to investigate different approaches to indeterminate thyroid nodules across different countries worldwide
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Rate of malignancy | 36 months
  Number of cancers over the total patients submitted to thyroidectomy for indeterminate thyroid nodules
Surgical approach to indeterminate thyroid nodules | 36 months
  Number of lobectomies over the total patients submitted to thyroidectomy for indeterminate thyroid nodules

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Cagliari, Cagliari, CA, Italy

IPD SHARING:
Plan to Share IPD: Undecided